CLINICAL TRIAL: NCT02755415
Title: Clinical Applicability of Robot-assisted Gait Training System in Acute Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH105-REC1-037
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Stroke
Keywords: Rehabilitation; Robotic; Gait; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Static Standing Table Training (Active Comparator): Patients in this group will receive standard hospital based rehabilitation as well as static standing table training
  Interventions: Other: Static Standing Table
- Robotic Gait Training (Experimental): Patients in this group will receive standard hospital based rehabilitation as well as robot-assisted gait rehabilitation training
  Interventions: Device: HIWIN Robotic Gait Training System

INTERVENTIONS:
Device: HIWIN Robotic Gait Training System — HIWIN Robotic Gait Training System is an automatic training system that combines weight-bearing standing, repetitive stepping and gait training
  Arms: Robotic Gait Training
Other: Static Standing Table — As part of the standard hospital rehabilitation, static standing table allows patient to be in a fully supported standing position
  Arms: Static Standing Table Training

SUMMARY:
Investigation of the clinical feasibility and efficacy of a newly developed robot-assisted gait training system for acute stroke survivors. It is anticipated that robot-assisted gait rehabilitation will achieve significantly better gait and quality of life outcomes than the standing table rehabilitation.

DETAILED DESCRIPTION:
Stroke is not only the second leading cause of mortality in Taiwan, it is also the primary cause of long-term physical and psychological disabilities in our society. Array of reasons have been suggested to be an obstacle for stroke patients to receive adequate physical rehabilitation, including the lack of physical capacity, severe neurological deficits or the loss of strength. Given the critical importance of high-intensity and high-repetitiveness of early rehabilitation for stroke patients in achieving sustainable long term outcomes, robot-assisted gait rehabilitation devices have gained great interest in the last decade and is slowly becoming part of the clinical rehabilitation program for stroke patients. However, despite the growing interest and the significant resources invested for the development of robot-assisted rehabilitation devices, there still lacks empirical evidence of its clinical applicability for stroke patients. Moreover, available evidence to date have mostly focused on sub-acute and chronic stroke patients and investigation in acute stroke population, especially in those with complete incapacitation for ambulation, is sparse. It is therefore the aim of the proposed project to fulfil this significant gap in our clinical knowledge by comparatively investigate the clinical applicability of a recently developed HIWIN Robotic Gait Training System (MRG-P100) against the traditional rehabilitation program with an emphasis on the determination of psychological and functional capacity recovery status in acute stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 20-80 years;
* Diagnosis of first, single unilateral cortical-subcortical acute stroke verified by brain imaging;
* Paresis of a lower limb;
* Ability to walk for only a few meters either with or without aid.

Exclusion Criteria:

* Deemed by a physician to be medically unstable;
* Other prior musculoskeletal conditions that affected gait capacity;
* Co-existence of other neurological diseases;
* Cognitive impairments that would impact on the safe participation in the study (MMSE<23)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 15-20 minutes
  The Berg Balance Scale (or BBS) is a widely used clinical test of a person's static and dynamic balance abilities and is generally considered to be the gold standard for clinical practice

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 10-15 minutes
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The questionnaire has been used in many settings, including research and clinical activities, and has been used in the diagnosis of sleep disorders
EuroQol five dimensions questionnaire (EQ-5D) | 10-15 minutes
  EuroQol five dimensions questionnaire (EQ-5D) is a standardized instrument for measuring generic health status.
Resting muscle tone | 10 minutes
  A device developed by Myoton Technology (Myoton AS, Estonia) will be used to determine the resting muscle tone (oscillation frequency [Hz]) of the tibialis anterior muscle, gastrocnemius muscle, rectus femoris muscle and biceps femoris muscle.
Resting muscle elasticity | 10 minutes
  A device developed by Myoton Technology (Myoton AS, Estonia) will be used to determine the resting muscle elasticity (Oscillation stiffness [N/m]) of the tibialis anterior muscle, gastrocnemius muscle, rectus femoris muscle and biceps femoris muscle.
Six minute walk test | 6 minutes
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway.
Beck's depression Inventory | 7-10 minutes
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will remain confidential and accessible to only the approved researchers